CLINICAL TRIAL: NCT04688138
Title: Predictive Value of Gut Microbiota and Serum Markers for Cognitive Impairment and Poor Prognosis After Ischemic Stroke: A Multiple Center Cohort Study
Brief Title: Gut Microbiota and Serum Markers for Cognitive Impairment and Poor Prognosis After Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangdong 999 Brain Hospital (Other); Zhujiang Hospital (Other); First Affiliated Hospital of Jinan University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2020-169
Record Dates: First submitted 2020-12-11; First posted 2020-12-29 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; cognitive impairment; gut microbiota
MeSH Terms: conditions — Ischemic Stroke; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasm; Faeces ;Oral swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ischemic stroke: Patients with ischemic stroke within 7 days of onset

SUMMARY:
Post-stroke cognitive impairment(PSCI) is one of the most important factors causing disabilities after stroke. Recent study found that gut microbiota plays a key role in neurological diseases. Two recent small sample studies reported gut dysbiosis in PSCI patients. In order to further verify the relationship between PSCI and gut microbiota and the predictive value of gut microbiota and serum markers for cognitive impairment and poor prognosis after ischemic stroke. The study intended to collect stool specimens of patients with acute ischemic stroke and assess their cognitive psychological state, and to establish a prospective multi-center follow-up cohort to explore the correlation between the dynamic changes of intestinal flora in patients with stroke and PSCI and poor prognosis of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for acute ischemic stroke;
* Aged between 18-75;
* Onset within 7 days;
* Sign informed consent and agree to provide relevant medical history data and biological specimens.

Exclusion Criteria:

* Patients diagnosed with TIA
* Severe disturbance of consciousness (NIHSS consciousness score > 1)
* Previous severe mental disorders and dementia (AD8 score ≥ 2)
* History of cerebral hemorrhage or any stroke within 12 months;
* Serious systemic diseases including malignant tumors
* Patients with aphasia and unable to cooperate to complete the Montreal Cognitive Assessment (MoCA)
* ALT or AST greater than 2 times the upper limit of normal value or severe liver disease;
* GFR less than 30mL/min/1.72m2 or severe kidney disease
* Alcohol abused, drug use and chemical poisoning history (such as pesticide poisoning)
* Patients with previous history of gastrointestinal tract or confirmed during hospitalization
* Patients who could not collect stool samples within 4 days after admission.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke within 7 days of onset
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | 7 days after admission
  A cognitive function screening test ranged 0-30, higher scores mean better cognitive function
Mini-Mental State Examination | 3 months after discharge
  A cognitive function screening test ranged 0-30, higher scores mean better cognitive function
Mini-Mental State Examination | 6 months after discharge
  A cognitive function screening test ranged 0-30, higher scores mean better cognitive function
Montreal Cognitive Assessment | 7 days after admission
  A cognitive function screening test ranged 0-30, higher scores mean better cognitive function
Montreal Cognitive Assessment | 3 months after discharge
  A cognitive function screening test ranged 0-30, higher scores mean better cognitive function
Montreal Cognitive Assessment | 6 months after discharge
  A cognitive function screening test ranged 0-30, higher scores mean better cognitive function
Gut microbiota | 2 days after admission
  Results of fecal bacteria by 16s RNA sequencing
Gut microbiota | 3 months after discharge
  Results of fecal bacteria by 16s RNA sequencing

SECONDARY OUTCOMES:
Modified Rankin Scale(mRS) | 7 days after admission
  A neurological function score scale ranged 0-6, higher scores mean worse neurological outcome
Modified Rankin Scale(mRS) | 3 months after discharge
  A neurological function score scale ranged 0-6, higher scores mean worse neurological outcome
Modified Rankin Scale(mRS) | 6 months after discharge
  A neurological function score scale ranged 0-6, higher scores mean worse neurological outcome
Modified Rankin Scale(mRS) | 12 months after discharge
  A neurological function score scale ranged 0-6, higher scores mean worse neurological outcome
National Institute of Health stroke scale(NIHSS) | Day 1 of admission
  Neurological function score scale, ranged 0-42, higher scores mean more severe neurological deficit
National Institute of Health stroke scale(NIHSS) | Day 7 of admission
  Neurological function score scale, ranged 0-42, higher scores mean more severe neurological deficit
National Institute of Health stroke scale(NIHSS) | 3 months after discharge
  Neurological function score scale, ranged 0-42, higher scores mean more severe neurological deficit
National Institute of Health stroke scale(NIHSS) | 6 months after discharge
  Neurological function score scale, ranged 0-42, higher scores mean more severe neurological deficit
Short chain fatty acids | 2 days after admission
  A metabolites of gut microbiota from stool, detected by gas chromatography-mass spectrometry (GC-MS) combined technique
Short chain fatty acids | 3 months after discharge
  A metabolites of gut microbiota from stool, detected by gas chromatography-mass spectrometry (GC-MS) combined technique
Trimethylamine-N-Oxide | 2 days after admission
  A metabolites of gut microbiota in plasm, quantified by stable isotope dilution liquid chromatography tandem mass spectrometry
Trimethylamine-N-Oxide | 3 months after discharge
  A metabolites of gut microbiota in plasm, quantified by stable isotope dilution liquid chromatography tandem mass spectrometry
Untargeted Metabolomics | 2 days after admission
  Untargeted metabolomics refers to using gas chromatography-mass spectrometry (GC-MS) combined technique, without bias detection of all small molecule metabolites in plasma (mainly the relative molecular weight of 1000 Da endogenous small molecule compounds) levels.
Untargeted Metabolomics | 3 months after discharge
  Untargeted metabolomics refers to using gas chromatography-mass spectrometry (GC-MS) combined technique, without bias detection of all small molecule metabolites in plasma (mainly the relative molecular weight of 1000 Da endogenous small molecule compounds) levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, NanFang Hospital, Southern Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ren Y, Liang J, Li X, Deng Y, Cheng S, Wu Q, Song W, He Y, Zhu J, Zhang X, Zhou H, Yin J. Association between oral microbial dysbiosis and poor functional outcomes in stroke-associated pneumonia patients. BMC Microbiol. 2023 Oct 24;23(1):305. doi: 10.1186/s12866-023-03057-8. PMID 37875813